CLINICAL TRIAL: NCT00801021
Title: Treatment and/or Prevention of Urinary Tract Infections
Acronym: UTI
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biomedical Development Corporation (Industry)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Baylor College of Medicine (Other)
Responsible Party: Barbara Wells Trautner, M.D., Ph.D., Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: H-23281; 1R41DK082089-01 (NIH)
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2010-03-08 (Estimated); Status verified 2009-11

CONDITIONS: Cystitis; Urinary Tract Infections
Keywords: Cystitis; Urinary Tract Infections
MeSH Terms: conditions — Cystitis; Urinary Tract Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Frio Oral Rinse (Experimental): Prescription Mouth Rinse
  Interventions: Drug: Frio Mouth Rinse

INTERVENTIONS:
Drug: Frio Mouth Rinse — Rinse with 15ml twice daily then expectorate
  Other Names: Prescription Mouth Rinse

SUMMARY:
The purpose of the study is to determine the effect of an investigational oral rinse in reducing uropathogens and treating uncomplicated urinary tract infections.

DETAILED DESCRIPTION:
A 7-day treatment with a 28-day follow up has been designed as a "before and after" assessment of the clinical signs and symptoms of an uncomplicated urinary tract infection and the reduction/eradication of urinary pathogens. Enrollment is targeted to achieving 20 evaluable subjects by the end of the study. After enrolling in the trial at Day 0 (first day of dosing), participants will report back to the study site at Days 3, 7, and 28. At Day 3 or any time thereafter, worsening of symptoms and/or increases in quantitative bacteria counts will result in removal from the trial and prescription of a rescue medication, which will be selected based on microbial susceptibility testing.

ELIGIBILITY:
Inclusion Criteria:

1. Non-pregnant adult females;
2. 18 years of age or older;
3. Clinical signs with one or more symptoms of a UTI (e.g., dysuria, frequency, urgency, suprapubic pain) with onset of symptoms < 72 hours prior to study entry;
4. One positive dipstick urine test positive either for leukocyte esterase or nitrates or have a urinalysis with > 5 wbc/hpf.
5. A pre-treatment clean-catch midstream urine culture with ≥ 104 CFU/mL of a bacterial organism

Exclusion Criteria:

1. Males;
2. Women who are pregnant, nursing, or not using a medically accepted, effective method of birth control;
3. Three or more episodes of acute uncomplicated UTI in the past 12 months;
4. Known structural abnormality that would predispose the participant to reflux or urinary retention;
5. Patients with evidence of factors predisposing to the development of urinary tract infections, including calculi, stricture, primary renal disease (e.g., polycystic renal disease), or neurogenic bladder;
6. Patients with significant impaired immunity secondary to chemotherapy, oral corticosteroids, or HIV;
7. Patients with onset of symptoms > 72 hours prior to entry;
8. Patients with a temperature ≥ 100°F, flank pain, chills, or any other manifestations suggestive of upper urinary tract infection;
9. Patients with purported hypersensitivity to iodine;
10. Patients with history of thyroid disease;
11. Patients who received treatment with other antimicrobials within 48 hours prior to entry;
12. Any significant medical or psychiatric condition that would render examination difficult or invalid or prevent the subject from active study participation; inability to use an oral rinse;
13. Use of concomitant medication that, in the opinion of the Study Directors, might interfere with the outcome of the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-12; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is the reduction of the baseline pathogen at the Days 7 to 10 "Test of Cure" visit. | 7 to 10 Days

SECONDARY OUTCOMES:
The secondary efficacy endpoint of microbiological evaluation classified into four categories (i.e., Eradication, Persistence, Superinfection, and New Infection) | 28-35 Days

CONTACTS AND LOCATIONS:
Overall Officials: Barbara W. Trautner, M.D., Ph.D., Principal Investigator — Baylor College of Medicine
Locations (1):
- Ben Taub General Hospital, Houston, Texas, United States